CLINICAL TRIAL: NCT01609478
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 12-week Treatment, Parallel-group Study to Assess the Efficacy, Safety and Pharmacokinetics of Indacaterol Acetate (75 and 150 µg o.d.) in Patients With Persistent Asthma
Brief Title: Efficacy, Safety and Pharmacokinetics of Indacaterol Acetate in Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQMF149E2203; 2012-000520-18 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-06-01 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — indacaterol; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- indacaterol acetate 75 µg (Experimental): indacaterol acetate 75 µg od delivered via Concept 1 inhaler
  Background therapy: mometasone furoate 200 mcg od
  Interventions: Drug: indacaterol; Drug: mometasone furoate
- indacaterol acetate 150 µg (Experimental): indacaterol acetate 150 µg od delivered via Concept 1 inhaler
  Background therapy: mometasone furoate 200 mcg od
  Interventions: Drug: indacaterol; Drug: mometasone furoate
- placebo (Placebo Comparator): placebo delivered via Concept 1 inhaler
  Background therapy: mometasone furoate 200 mcg od
  Interventions: Drug: placebo; Drug: mometasone furoate

INTERVENTIONS:
Drug: indacaterol — indacaterol acetate 75 µg or indacaterol acetate 150 µg delivered via Concept 1 inhaler
  Arms: indacaterol acetate 150 µg; indacaterol acetate 75 µg
Drug: placebo — placebo delivered via Concept 1 inhaler
  Arms: placebo
Drug: mometasone furoate — via Twisthaler inhaler

SUMMARY:
To provide the efficacy, safety and pharmacokinetics of indacaterol acetate in patients with persistent asthma to support dose selection of indacaterol in fixed dose combination QMF149.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent asthma, diagnosed according to GINA 2010 guideline and who additionally meet the following criteria:
* Patients who are receiving ICS treatment in a stable regimen for ≥ 4 weeks
* Patients with a pre-bronchodilator FEV1 value of ≥ 40% and ≤ 80% of predicted normal value
* Patients who demonstrate an increase of >= 12% and 200 mL in FEV1
* ACQ-5 score ≥ 1.5

Exclusion Criteria:

* Patients who are current smokers or have a smoking history of greater than 10 pack years (defined as the number of packs of 20 cigarettes smoked per day multiplied by number of years the patient smoked).
* Patients with chronic lung disease, including COPD, pulmonary tuberculosis, bronchiectasis, sarcoidosis, interstitial lung disease and cystic fibrosis.
* Patients with any chronic conditions affecting the respiratory tract (e.g., chronic sinusitis) which in the opinion of the investigator may interfere with the study evaluation or optimal participation in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (84):
- Bulgaria (9):
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Lovech
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (12):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Downsview, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Grimsby, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Woodstock, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Saint Romuald, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
- Germany (10):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Wiesloch
- Japan (22):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Ako-shi, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Beppu, Oita Prefecture
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Cyuo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Machida-shi, Tokyo-To
  - Novartis Investigative Site, Ōta-ku, Tokyo-To
  - Novartis Investigative Site, Yonezawa, Yamagata
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard-Geleen
- Poland (10):
  - Novartis Investigative Site, Gdansk, Poland
  - Novartis Investigative Site, Krakow, Poland
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bieńkówka
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Żnin
- Slovakia (15):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
  - Novartis Investigative Site, Dunajská Streda
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Liptovský Hrádok
  - Novartis Investigative Site, Liptovský Mikuláš
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Spisská Nová Ves
  - Novartis Investigative Site, Topoľčany
  - Novartis Investigative Site, Vyšné Hágy
- South Korea (4):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Started | 111 | 108 | 116
Full Analysis Set (FAS) | 110 | 108 | 115
Completed | 104 | 106 | 107
Not Completed | 7 | 2 | 9
Not completed — Adverse Event | 3 | 1 | 5
Not completed — Protocol Deviation | 0 | 1 | 1
Not completed — Non-Compliance with study treatment | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo | Total
Number analyzed (Participants) | 111 | 108 | 116 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (14.74) | 48.1 (13.53) | 49.8 (12.96) | 49.6 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 61 | 180
  Male | 52 | 48 | 55 | 155

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) After 12 Weeks (Day 85)
Description: Forced Expiratory Volume in 1 second (FEV1) was measured via spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose after 12 weeks (Day 85)
Time Frame: after 12 weeks (Day 85)
Population: The Full Analysis Set (FAS) included all randomized who received at least one dose of study drug with available data for analysis. Participants from FAS were considered for this analysis, however for a given time point participants analyzed had a value at such timepoint.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 107 | 104 | 111
Liters | 2.190 (0.0283) | 2.216 (0.0281) | 2.110 (0.0275)

2. Secondary Outcome: Asthma Control Questionnaire 5 (ACQ-5) After 12 Weeks (Day 85)
Description: The Asthma Control Questionnaire (ACQ-5) is a validated questionnaire consisting of 5 items for the assessment of asthma symptom which are night symptom, morning symptom, limitation for the activities, shortness of breath, and wheeze. The ACQ-5 score is the mean of the 5 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). A negative change in score indicates improvement in symptoms. MIXED model: Change from baseline in ACQ-5 = treatment + gender + baseline ACQ-5 score + age + level of asthma control + region + center (region) + error. Center is included as a random effect nested within region.
Time Frame: aftert 12 weeks (Day 85)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 103 | 104 | 108
Units on a Scale | 1.31 (0.094) | 1.42 (0.093) | 1.32 (0.092)

3. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) After 2 Weeks (Day 15), 4 Weeks (Day 29), and 8 Weeks (Day 57) of Treatment.
Description: Forced Expiratory Volume in 1 second (FEV1) was measured via spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose after 2 weeks (Day 15), 4 weeks (Day 29), and 8 weeks (Day 57) of treatment.
Time Frame: Day 15, Day 29 and Day 57
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 107 | 104 | 111
Liters
  Day 15 | 2.169 (0.0259) | 2.198 (0.0260) | 2.069 (0.0253)
  Day 29 | 2.180 (0.0274) | 2.196 (0.0276) | 2.057 (0.0266)
  Day 57 | 2.180 (0.0281) | 2.227 (0.0281) | 2.099 (0.0273)

4. Secondary Outcome: Forced Vital Capacity (FVC) on Day 1, Day 2, Day 14, Day 15, Day 84, Day 85 at All Time Points
Description: Forced Vital Capacity (FVC) was measured via spirometry conducted according to internationally accepted standards. FVC is measured on Day 1, Day 2, Day 14, Day 15, Day 84, Day 85 at all time points
Time Frame: Day 1, Day 2, Day 14, Day 15, Day 84, Day 85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
liters
  Day 1 / 5 min post-dose (n=107,105,111) | 3.342 (0.0198) | 3.338 (0.0198) | 3.235 (0.0190)
  Day 1 / 15 min post-dose (n=107,105,111) | 3.372 (0.0240) | 3.348 (0.0241) | 3.238 (0.0232)
  Day 1 / 30 min post-dose (n=107,104,111) | 3.378 (0.0236) | 3.367 (0.0236) | 3.239 (0.0227)
  Day 1 / 1 hr post-dose (n=107,104,111) | 3.356 (0.0237) | 3.333 (0.0239) | 3.241 (0.0229)
  Day 1 / 2 hr post-dose (n=106,104,111) | 3.366 (0.0256) | 3.367 (0.0258) | 3.268 (0.0247)
  Day 1 / 4 hr post-dose (n=107,101,111) | 3.346 (0.0304) | 3.342 (0.0307) | 3.238 (0.0290)
  Day 1 / 6 hr post-dose (n=24,24,26) | 3.299 (0.0545) | 3.345 (0.0507) | 3.280 (0.0509)
  Day 2 / 23 hr 10min post-dose (n=107,104,110) | 3.314 (0.0282) | 3.303 (0.0290) | 3.254 (0.0279)
  Day 2 / 23 hr 45min post-dose (n=107,104,111) | 3.313 (0.0309) | 3.341 (0.0314) | 3.269 (0.0297)
  Day 14 / 5 min post-dose (n=107,105,111) | 3.404 (0.0327) | 3.364 (0.0332) | 3.212 (0.0326)
  Day 14 / 15 min post-dose (n=107,105,111) | 3.397 (0.0340) | 3.377 (0.0343) | 3.213 (0.0336)
  Day 14 / 30 min post-dose (n=107,104,111) | 3.412 (0.0341) | 3.389 (0.0345) | 3.246 (0.0336)
  Day 14 / 1 hr post-dose (n=107,104,111) | 3.408 (0.0324) | 3.379 (0.0327) | 3.206 (0.0319)
  Day 14 / 2 hr post-dose (n=106,104,111) | 3.402 (0.0325) | 3.395 (0.0329) | 3.207 (0.0323)
  Day 14 / 4 hr post-dose (n=107,101,111) | 3.368 (0.0329) | 3.338 (0.0336) | 3.217 (0.0323)
  Day 14 / 6 hr post-dose (n=24,24,26) | 3.332 (0.0620) | 3.426 (0.0584) | 3.257 (0.0602)
  Day 15 / 23 hr 10min post-dose (n=107,104,110) | 3.324 (0.0298) | 3.311 (0.0302) | 3.237 (0.0294)
  Day 15 / 23 hr 45min post-dose (n=107,104,111) | 3.347 (0.0307) | 3.313 (0.0311) | 3.260 (0.0301)
  Day 84 / 5 min post-dose (n=107,105,111) | 3.381 (0.0331) | 3.374 (0.0335) | 3.263 (0.0331)
  Day 84 / 15 min post-dose (n=107,105,111) | 3.393 (0.0353) | 3.392 (0.0355) | 3.275 (0.0351)
  Day 84 / 30 min post-dose (n=107,104,111) | 3.424 (0.0350) | 3.399 (0.0352) | 3.282 (0.0349)
  Day 84 / 1hr post-dose (n=107,104,111) | 3.394 (0.0339) | 3.393 (0.0346) | 3.262 (0.0336)
  Day 84 / 2 hr post-dose (n=106,104,111) | 3.413 (0.0334) | 3.382 (0.0335) | 3.292 (0.0332)
  Day 84 / 4 hr post-dose (n=106,101,111) | 3.346 (0.0350) | 3.363 (0.0356) | 3.257 (0.0349)
  Day 85 / 23 hr 10min post-dose (n=107,104,110) | 3.350 (0.0342) | 3.300 (0.0347) | 3.287 (0.0339)
  Day 85 / 23 hr 45min post-dose (n=107,104,111) | 3.343 (0.0367) | 3.321 (0.0368) | 3.294 (0.0360)

5. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)/ Forced Vital Capacity (FVC) on Day 1, Day 2, Day 14, Day 15, Day 84, Day 85
Description: Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) was measured via spirometry conducted according to internationally accepted standards.
Time Frame: Day 1, Day 2, Day 14, Day 15, Day 84, Day 85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
ratio
  Day 1 / 5 min post-dose (n=107,105,111) | 65.608 (0.3659) | 66.049 (0.3641) | 63.461 (0.3508)
  Day 1 / 15 min post-dose (n=107,105,111) | 65.602 (0.3854) | 67.039 (0.3898) | 63.537 (0.3759)
  Day 1 / 30 min post-dose (n=107,104,111) | 65.738 (0.4626) | 67.189 (0.4607) | 63.767 (0.4454)
  Day 1 / 1 hr post-dose (n=107,104,111) | 66.089 (0.4465) | 67.620 (0.4485) | 63.744 (0.4298)
  Day 1 / 2 hr post-dose (n=106,104,111) | 66.607 (0.4705) | 67.824 (0.4727) | 64.141 (0.4534)
  Day 1 / 4 hr post-dose (n=107,101,111) | 66.094 (0.5098) | 67.968 (0.5137) | 64.212 (0.4871)
  Day 1 / 6 hr post-dose (n=24,24,26) | 64.716 (0.9815) | 68.846 (0.9220) | 63.773 (0.9135)
  Day 2 / 23 hr 10min post-dose (n=107,104,110) | 65.465 (0.5112) | 66.942 (0.5197) | 63.822 (0.5006)
  Day 2 / 23 hr 45min post-dose (n=107,104,111) | 65.809 (0.5299) | 66.791 (0.5323) | 63.741 (0.5057)
  Day 14 / 5 min post-dose (n=107,105,111) | 66.548 (0.5102) | 67.366 (0.5172) | 64.362 (0.5075)
  Day 14 / 15 min post-dose (n=107,105,111) | 67.187 (0.5042) | 67.577 (0.5093) | 64.702 (0.4986)
  Day 14 / 30 min post-dose (n=107,104,111) | 67.024 (0.5601) | 67.765 (0.5633) | 64.192 (0.5476)
  Day 14 / 1 hr post-dose (n=107,104,111) | 67.100 (0.5446) | 68.262 (0.5476) | 64.383 (0.5327)
  Day 14 / 2 hr post-dose (n=106,104,111) | 67.538 (0.5486) | 68.397 (0.5540) | 64.617 (0.5431)
  Day 14 / 4 hr post-dose (n=107,101,111) | 66.866 (0.5763) | 68.044 (0.5871) | 64.426 (0.5632)
  Day 14 / 6 hr post-dose (n=24,24,26) | 64.792 (1.0246) | 67.346 (0.9676) | 64.167 (0.9834)
  Day 15 / 23 hr 10min post-dose (n=107,104,110) | 65.436 (0.5564) | 65.930 (0.5597) | 64.027 (0.5455)
  Day 15 / 23 hr 45min post-dose (n=107,104,111) | 65.606 (0.5871) | 66.435 (0.5887) | 63.726 (0.5729)
  Day 84 / 5 min post-dose (n=107,105,111) | 67.040 (0.5442) | 67.762 (0.5498) | 64.850 (0.5422)
  Day 84 / 15 min post-dose (n=107,105,111) | 67.162 (0.5671) | 67.907 (0.5719) | 65.074 (0.5646)
  Day 84 / 30 min post-dose (n=107,104,111) | 66.936 (0.6017) | 67.865 (0.6031) | 64.848 (0.5966)
  Day 84 / 1hr post-dose (n=107,104,111) | 3.394 (0.0339) | 3.393 (0.0346) | 3.262 (0.0336)
  Day 84 / 2 hr post-dose (n=106,104,111) | 3.413 (0.0334) | 3.382 (0.0335) | 3.292 (0.0332)
  Day 84 / 4 hr post-dose (n=106,101,111) | 3.346 (0.0350) | 3.363 (0.0356) | 3.257 (0.0349)
  Day 85 / 23 hr 10min post-dose (n=107,104,110) | 3.350 (0.0342) | 3.300 (0.0347) | 3.287 (0.0339)
  Day 85 / 23 hr 45min post-dose (n=107,104,111) | 3.343 (0.0367) | 3.321 (0.0368) | 3.294 (0.0360)

6. Secondary Outcome: Forced Expiratory Flow (FEF 25-75% )on Day 1, Day 2, Day 14, Day 15, Day 84, Day 85
Description: Forced Expiratory Flow (FEF 25-75%) was measured via spirometry conducted according to internationally accepted standards.
Time Frame: Day 1, Day 2, Day 14, Day 15, Day 84, Day 85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
liters/second
  Day 1 / 5 min post-dose (n=107,105,111) | 1.420 (0.0237) | 1.485 (0.0235) | 1.295 (0.0226)
  Day 1 / 15 min post-dose (n=107,105,111) | 1.449 (0.0254) | 1.563 (0.0256) | 1.295 (0.0247)
  Day 1 / 30 min post-dose (n=107,104,111) | 1.467 (0.0290) | 1.568 (0.0290) | 1.310 (0.0280)
  Day 1 / 1 hr post-dose (n=107,104,111) | 1.471 (0.0307) | 1.594 (0.0309) | 1.297 (0.0296)
  Day 1 / 2 hr post-dose (n=106,104,111) | 1.508 (0.0307) | 1.632 (0.0310) | 1.348 (0.0297)
  Day 1 / 4 hr post-dose (n=107,101,111) | 1.479 (0.0327) | 1.625 (0.0331) | 1.329 (0.0313)
  Day 1 / 6 hr post-dose (n=24,24,26) | 1.364 (0.0889) | 1.620 (0.0840) | 1.332 (0.0832)
  Day 2 / 23 hr 10min post-dose (n=107,104,110) | 1.407 (0.0322) | 1.520 (0.0328) | 1.310 (0.0315)
  Day 2 / 23 hr 45min post-dose (n=107,104,111) | 1.436 (0.0399) | 1.524 (0.0401) | 1.326 (0.0382)
  Day 14 / 5 min post-dose (n=107,105,111) | 1.505 (0.0350) | 1.571 (0.0354) | 1.318 (0.0348)
  Day 14 / 15 min post-dose (n=107,105,111) | 1.540 (0.0366) | 1.597 (0.0370) | 1.351 (0.0362)
  Day 14 / 30 min post-dose (n=107,104,111) | 1.532 (0.0383) | 1.607 (0.0386) | 1.336 (0.0376)
  Day 14 / 1 hr post-dose (n=107,104,111) | 1.569 (0.0400) | 1.664 (0.0402) | 1.343 (0.0391)
  Day 14 / 2 hr post-dose (n=106,104,111) | 1.551 (0.0380) | 1.676 (0.0385) | 1.338 (0.0379)
  Day 14 / 4 hr post-dose (n=107,101,111) | 1.526 (0.0434) | 1.628 (0.0445) | 1.339 (0.0426)
  Day 14 / 6 hr post-dose (n=24,24,26) | 1.370 (0.0843) | 1.519 (0.0792) | 1.363 (0.0808)
  Day 15 / 23 hr 10min post-dose (n=107,104,110) | 1.421 (0.0383) | 1.442 (0.0386) | 1.315 (0.0377)
  Day 15 / 23 hr 45min post-dose (n=107,104,111) | 1.430 (0.0431) | 1.492 (0.0431) | 1.319 (0.0420)
  Day 84 / 5 min post-dose (n=107,105,111) | 1.535 (0.0391) | 1.627 (0.0394) | 1.363 (0.0390)
  Day 84 / 15 min post-dose (n=107,105,111) | 1.530 (0.0393) | 1.675 (0.0396) | 1.372 (0.0392)
  Day 84 / 30 min post-dose (n=107,104,111) | 1.548 (0.0412) | 10659 (0.0414) | 1.368 (0.0411)
  Day 84 / 1hr post-dose (n=107,104,111) | 1.578 (0.0408) | 1.687 (0.0415) | 1.404 (0.0404)
  Day 84 / 2 hr post-dose (n=106,104,111) | 1.571 (0.0409) | 1.704 (0.0411) | 1.382 (0.0409)
  Day 84 / 4 hr post-dose (n=106,101,111) | 1.548 (0.0398) | 1.648 (0.0405) | 1.350 (0.397)
  Day 85 / 23 hr 10min post-dose (n=107,104,110) | 1.437 (0.0378) | 1.507 (0.0380) | 1.328 (0.0373)
  Day 85 / 23 hr 45min post-dose (n=107,104,111) | 1.476 (0.0428) | 1.496 (0.0427) | 1.378 (0.0418)

7. Secondary Outcome: Standardized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) at (5 Min - 4 h), (5 Min - 1 h) (1 h - 4 h) Measured on Day 1, 2 Weeks (Day 14)&12 Weeks (Day 84)
Description: Forced Expiratory Volume in 1 second (FEV1)/Area Under the Curve(AUC) was measured via spirometry conducted according to internationally accepted standards.FEV1 AUC(5 min - 4 h), (5 min - 1 h) and (1 h - 4 h) are measured at Day 1, 2 Weeks (Day 14) and 12 Weeks (Day84) and defined as average of FEV1 at specified timepoints above.
Time Frame: Day 1, 2 Weeks, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
Liters
  Day 1 (5min-4h) (n=107,105,111) | 2.209 (0.0170) | 2.274 (0.0169) | 2.077 (0.0163)
  Day 1 (5min-1h) (n=107,105,111) | 2.198 (0.0165) | 2.253 (0.0164) | 2.059 (0.0158)
  Day 1 (1h-4h) (n=107,104,111) | 2.212 (0.0182) | 2.284 (0.0183) | 2.082 (0.0175)
  Day 14 (5min-4h) (n=107,105,111) | 2.265 (0.0244) | 2.313 (0.0246) | 2.074 (0.0240)
  Day 14 (5min-1h) (n=107,105,111) | 2.267 (0.0245) | 2.299 (0.0246) | 2.069 (0.0241)
  Day 14 (1h-4h) (n=107,104,111) | 2.262 (0.0247) | 2.318 (0.0250) | 2.066 (0.0244)
  Day 84 (5min-4h) (n=107,105,111) | 2.264 (0.0259) | 2.322 (0.0260) | 2.132 (0.0257)
  Day 84 (5min-1h) (n=107,105,111) | 2.265 (0.0271) | 2.321 (0.0272) | 2.119 (0.0270)
  Day 84 (1h-4h) (n=107,104,111) | 2.263 (0.0258) | 2.322 (0.0260) | 2.130 (0.0257)

8. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) at Day 1, 2 Weeks (Day 14), 12 Weeks (Day 84)
Description: Peak Forced Expiratory Volume in 1 second (FEV1) was measured via spirometry conducted according to internationally accepted standards. Peak FEV1 is defined as the maximum FEV1 during the first 4 h post morning dosing at Day 1, 2Weeks and 12 Weeks.
Time Frame: Day 1, 2 weeks (Day 14), 12 weeks (Day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
liters
  Day 1 | 2.287 (0.0183) | 2.353 (0.0182) | 2.172 (0.0176)
  Day 14 | 2.345 (0.0252) | 2.387 (0.0254) | 2.165 (0.0248)
  Day 84 | 2.345 (0.0272) | 2.403 (0.0273) | 2.215 (0.0270)

9. Secondary Outcome: Asthma Control Questionnaire 5 (ACQ-5) After 4 Weeks (Day 29) and After 8 Weeks (Day 57) of Treatment
Description: The ACQ-5 is a validated questionnaire consisting of 5 items for the assessment of asthma symptom which are night symptom, morning symptom, limitation for the activities, shortness of breath, and wheeze. Each item is graded on a scale of 0-6 and the questions are equally weighted. The ACQ-5 score is the mean of the 5 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: after 4 weeks (Day 29) and after 8 weeks (Day 57)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
units on a scale
  Day 29 (n=103, 104, 108) | 1.43 (0.088) | 1.39 (0.088) | 1.55 (0.086)
  Day 57 (n= 103, 104, 108) | 1.42 (0.093) | 1.29 (0.093) | 1.46 (0.091)

10. Secondary Outcome: Morning and Evening Peak Expiratory Flow Rate (PEFR) Over 12 Weeks of Treatment. This is LS Mean of the Treatment Period.
Description: PEFR is measured with portable spirometer by participants every morning and evening at home.
Time Frame: baseline, 4weeks, 8 weeks and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
liters/second
  Morning Baseline - <4 weeks (n=104,100,109) | 326.98 (3.741) | 335.44 (3.842) | 307.68 (3.636)
  Evening baseline - <4 weeks (n=104,100,109) | 332.96 (3.477) | 345.99 (3.587) | 312.42 (3.545)
  Morning 4 weeks - <8 weeks (n=104,100,109) | 328.45 (4.374) | 338.23 (4.466) | 315.60 (4.248)
  Evening 4 weeks - <8 weeks (n=104,100,109) | 333.36 (4.221) | 344.63 (4.323) | 313.31 (4.284)
  Morning 8 weeks - <12 weeks (n=104,100,109) | 329.85 (4.699) | 334.83 (4.783) | 317.03 (4.559)
  Evening 8 weeks - <12 weeks (n=104,100,109) | 332.61 (4.628) | 342.40 (4.718) | 316.28 (4.677)

11. Secondary Outcome: The Usage of Rescue Medication (Short Acting β2-agonist) Over 12 Weeks of Treatment
Description: Participants record the number of puffs of rescue medication taken in the previous 12 hours in the morning and nighttime.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: number of puffs
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
number of puffs
  Mean daily number of puffs (n=105, 102, 105) | 1.08 (0.132) | 0.99 (0.136) | 1.31 (0.132)
  Mean Daytime number of puffs (n=103, 99, 100) | 0.54 (0.074) | 0.55 (0.077) | 0.73 (0.076)
  Mean nighttime number of puffs (n=104, 100, 107) | 0.55 (0.063) | 0.47 (0.065) | 0.64 (0.062)

12. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ(S)) After 4 Weeks (Day 29) and 12 Weeks (Day 85) of Treatment
Description: The AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments in asthma. Patients are asked to score each item on a 7-point scale based on the experience of last 2 weeks. The overall AQLQ score is the mean response to all 32 questions. Therefore, the possible highest score (better) would be 7 and the lowest (worse) would be 1. Changes in scores of 0.5 to 1.0 are considered clinically meaningful; 1.0 to 1.5 as moderate and > 1.5 as marked clinically important differences for any individual domain or for the overall summary score.
Time Frame: 4 Weeks, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
Units on a Scale
  Day 29 (n=103,104, 108) | 5.52 (0.082) | 5.48 (0.082) | 5.38 (0.080)
  Day 85 (n=103,104, 108) | 5.64 (0.088) | 5.47 (0.087) | 5.60 (0.086)

13. Secondary Outcome: Time to First Asthma Exacerbation (Mild, Moderate, Severe, Moderate or Severe and Any) Over the 12 Week Treatment Period
Description: Duration of treatment until first asthma exacerbation by severity of exacerbation. A severe asthma exacerbation is systemic corticosteroids (SCS) use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
weeks
  Moderate or Severe exacerbation | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.
  Any Asthma Exacerbation | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.
  Mild Asthma Exacerbation | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.
  Moderate Asthma Exacerbation | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.
  Severe Asthma Exacerbation | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.

14. Secondary Outcome: The Annual Rate of Asthma Exacerbations (Mild, Moderate, Severe, Moderate or Severe and Any) Over the 12 Week Treatment Period
Description: Annual incidence rate of asthma exacerbation by severity of exacerbation. The number of asthma exacerbation is used to calculate annual incidence rate. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations. Number of the asthma exacerbation will be analyzed by the negative binomial regression including treatment, history of asthma exacerbation in the 12 months prior to screening and region as factors and FEV1 prior to inhalation and FEV1 30 min post inhalation of salbutamol/albuterol (components of SABA reversibility) as covariates. The estimates are obtained from the model and so we cannot specify a formula.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: # of exacerbations
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
# of exacerbations
  Moderate or Severe Exacerbation | 0.315 [0.1184 to 0.8387] | 0.353 [0.1373 to 0.9053] | 0.352 [0.1406 to 0.8805]
  Any asthma exacerbation | 0.421 [0.1711 to 1.0358] | 0.569 [0.2389 to 1.3553] | 0.788 [0.3486 to 1.7827]
  Mild Asthma Exacerbation | 0.000 [0.0000 to NA] — upper limit infinity | 0.001 [0.0000 to NA] — upper limit infinity | 0.001 [0.000 to NA] — upper limit infinity
  Moderate Asthma Exacerbation | 0.225 [0.0790 to 0.6403] | 0.320 [0.1239 to 0.8251] | 0.274 [0.1017 to 0.7387]
  Severe Asthma Exacerbation | 0.000 [0.0000 to NA] — upper limit infinity | 0.000 [0.000 to NA] — upper limit infinity | 0.000 [0.000 to NA] — upper limit infinity

15. Secondary Outcome: Duration of Asthma Exacerbations (Mild, Moderate, Severe, Moderate or Severe and Any) Over the 12 Week Treatment Period
Description: Duration of asthma exacerbations by severity of exacerbation. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
days
  moderate or severe exacerbations | 0.7 (3.32) | 0.6 (2.50) | 0.8 (4.11)
  any asthma exacerbations | 1.0 (3.88) | 0.9 (3.62) | 1.3 (4.74)
  mild asthma exacerbations | 0.3 (2.11) | 0.4 (2.47) | 0.5 (2.54)
  moderate asthma exacerbations | 0.6 (3.26) | 0.6 (2.50) | 0.6 (3.53)
  Severe asthma exacerbations | 0.1 (0.67) | 0.0 (0.00) | 0.1 (1.59)

16. Secondary Outcome: The Percentage of Patients With at Least One Asthma Exacerbation (Mild, Moderate, Severe, Moderate or Severe and Any) Over the 12 Week Treatment Period
Description: The percentage of patients with at least one asthma exacerbation by severity of exacerbation. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 107 | 105 | 111
percentage of participants
  moderate or severe asthma exacerbations | 5.6 | 5.7 | 4.5
  any asthma exacerbations | 8.4 | 8.6 | 9.9
  mild asthma exacerbations | 2.8 | 3.8 | 5.4
  moderate asthma exacerbations | 4.7 | 5.7 | 4.5
  severe asthma exacerbations | 0.9 | 0.0 | 0.9

17. Secondary Outcome: Time to Permanent Study Discontinuation Due to Asthma Exacerbation Over the 12 Week Treatment Period
Description: Time to permanent study discontinuation due to asthma exacerbation. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
days | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median. | NA [NA to NA] — There were too few events to calculate the median.

18. Secondary Outcome: The Percentage of Patients Who Permanently Discontinued Study Due to Asthma Exacerbation Over the 12 Week Treatment Period
Description: The percentage of patients who permanently discontinued study due to asthma exacerbation. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 107 | 105 | 111
percentage of participants | 1.9 | 1.0 | 3.6

19. Secondary Outcome: Total Amounts (in Doses) of Systemic Corticosteroids Used to Treat Asthma Exacerbations Over the 12 Week Treatment Period
Description: Total amounts (in doses) of systemic corticosteroids (SCS) used to treat asthma exacerbations.SCS includes Intramuscular (IM), Intravenous (IV) and Oral. A severe asthma exacerbation is SCS use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 110 | 108 | 115
milligrams (mg)
  IIntramuscular - Triamcinolone Acetonide | NA (NA) — no participants in this treatment group took this SCS | 20 (NA) — SD cannot be calculated as there was only one value | 0 (NA) — no participants in this treatment group took this SCS
  Intravenous - Betamethasone | NA (NA) — no participants in this treatment group took this SCS | 4 (NA) — SD cannot be calculated as there was only one value | 4 (NA) — SD cannot be calculated as there was only one value
  Intravenous- Hydrocortisone | 500 (NA) — SD cannot be calculated as there was only one value | 100 (NA) — SD cannot be calculated as there was only one value | 200 (NA) — SD cannot be calculated as there was only one value
  Intravenous- Hydrocortisone NA Succinate | 300 (NA) — SD cannot be calculated as there was only one value | 500 (141.421) | NA (NA) — no participants in this treatment group took this SCS
  Intravenous- Methylprednisolone NA Succinate | 60 (28.284) | 80 (NA) — SD cannot be calculated as there was only one value | NA (NA) — no participants in this treatment group took this SCS
  Oral- Methylprednisolone | NA (NA) — no participants in this treatment group took this SCS | 32 (NA) — SD cannot be calculated as there was only one value | NA (NA) — no participants in this treatment group took this SCS
  Oral - Prednisolone | 60 (42.426) | 90 (NA) — SD cannot be calculated as there was only one value | 37.50 (24.749)
  Oral - Prednisone | 40 (NA) — SD cannot be calculated as there was only one value | 40 (0) | 100 (70.11)
  Oral - Prednisone equivalent dose | 102 (66.765) | 106.11 (104.055) | 58.61 (49.956)

20. Secondary Outcome: Plasma Indacaterol Concentrations at Day 1 and Day 14
Description: Maximum plasma concentration after drug administration (Cmax) was measured for indacaterol acetate 75 µg and indacaterol acetate 150 µg for Pharmacokinetic (PK) Subgroup
Time Frame: Day 1 and Day 14
Population: Pharmacokinetic (PK) profiling subgroup included all randomized patients who consented to participate in the additional PK assessment.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Indacaterol Acetate 75 µg | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 30 | 26
pg/ml
  Day 1 (n=21, 21) | 70.7 (29.1) | 164 (69.5)
  Day 14 (n=21, 21) | 129 (48.6) | 285 (108)

ADVERSE EVENTS:
Groups:
- Indacaterol Acetate 75 mcg: indacaterol acetate 75 µg od delivered via Concept 1 inhaler Background therapy: mometasone furoate 200 mcg od
- Indacaterol Acetate 150 mcg: indacaterol acetate 150 µg od delivered via Concept 1 inhaler Background therapy: mometasone furoate 200 mcg od
Arm/Group | Indacaterol Acetate 75 mcg | Indacaterol Acetate 150 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/110 | 0/108 | 2/115
Other Adverse Events (participants affected / at risk) | 19/110 | 20/108 | 28/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Acetate 75 mcg (N=110) | Indacaterol Acetate 150 mcg (N=108) | Placebo (N=115)
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Acetate 75 mcg (N=110) | Indacaterol Acetate 150 mcg (N=108) | Placebo (N=115)
NASOPHARYNGITIS (Infections and infestations) | 7 | 6 | 9
PHARYNGITIS (Infections and infestations) | 1 | 1 | 4
RHINITIS (Infections and infestations) | 0 | 3 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
HEADACHE (Nervous system disorders) | 5 | 2 | 4
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.